CLINICAL TRIAL: NCT02368054
Title: Hemodynamic Stability of Bupivacaine With and Without Adrenaline for Paracervical Block for Cervical Conization During General Anesthesia: A Randomized Controlled Double Blinded Study
Brief Title: Hemodynamic Stability of Bupivacaine With and Without Adrenaline for Paracervical Block for Cervical Conization
Acronym: HSBAPCB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Gunnar Helge Sjøen, Anesthesiologist, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 49024; 2014-004504-29 (EudraCT Number); 2014/1909/REK-vest (Other: Regional Ethical Comittee)
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Epinephrine; Bupivacaine; Stroke Volume; Cardiac Output; Heart Rate; Hemodynamics; Total Peripheral Resistance; Blood Pressure; Paracervical block; LiDCO; Adrenaline; Conization; PulsCO
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine-adrenaline (Active Comparator): Paracervical block. Bupivacaine 2,5 mg/ml Adrenaline 5 microg/ml; 20 ml
  Interventions: Drug: Bupivacaine; Drug: Adrenaline
- Bupivacaine (Active Comparator): Paracervical block. Bupivacaine 2,5 mg/ml; 20 ml
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Infiltration anesthesia
  Other Names: Marcain
Drug: Adrenaline — Infiltration anesthesia
  Other Names: Epinephrine
  Arms: Bupivacaine-adrenaline

SUMMARY:
Cervical conization is done for pre-cancer disease. The procedure is performed with local anesthesia and general anesthesia. Local anesthesia is given by paracervical block, and several different local anesthetics is being used including bupivacaine with and without adrenaline. Adrenaline might reduce local bleeding and reduce toxicity of bupivacaine by reducing absorption, but might affect cardiovascular function. This study will examine this effect.

DETAILED DESCRIPTION:
Most patients scheduled for cervical conization are healthy, young women. Some do this procedure with local anesthesia (paracervical block) and sedation, others general anesthesia combined with local anesthesia. Lidocaine with adrenaline is often used, but some uses longer acting substances like bupivacaine 2,5 mg/ml with adrenaline 5 microg/ml.

Adding of adrenaline prolongs the effect of anesthesia and the effect is probably strongest for short-acting local anesthetics. Adrenaline may delay absorption of local anesthetics avoiding toxic plasma concentrations and reduce local bleeding. Injection of local anesthetics with adrenaline may affect haemodynamic stability.

Para-cervical block has been used for analgesia in first stage of labor, but may give foetal bradycardia in 3-4 % and may affect the cardiotocogram in 10-12%. This effect is observed with bupivacaine and the less toxic levobupivacaine. Because of fear for complications and foetal injury this block has been replaced by more effective and safer methods like epidural and spinal anesthesia.

In gynecological practice the para-cervical block is still used for termination of pregnancy, cervical conization and for instrumentation of uterus.

We have observed affection of hemodynamic stability when using local anesthetics with adrenaline in nasal mucosa and during cervical conization. Some patients may experience increase or decrease in blood pressure and heart rate with a duration of 3-5 minutes.

Kerkkamp and coworkers have observed an 64% increase in cardiac output when using bupivacaine with adrenaline 100 microg epidurally but de Leeuw et al find an effect of less than 10% change in cardiac output during combined psoas compartment and ischiadic-block. We have performed a non-randomized, non-blinded pilot-study showing a 86% increase in systolic blood pressure and 65% increase in cardiac output after para-cervical block with bupivacaine 50 mg and adrenaline 100 microg. We want to confirm these results by doing a randomized, blinded study.

Most day-surgical patients are classified as ASA (American Society of Anesthesiologists) grade 1-2, and the complication rates are low. Still we may experience cardiovascular events during anesthesia with patients considered without cardiovascular diseases. Hemodynamic stability during anesthesia is a goal for all patients.

LiDCOplus (Lithium Dilution Cardiac Output) is a minimal invasive hemodynamic monitor for measuring cardiac output (CO) and systemic resistance (SVR). It uses two algorithms. PulseCO is an analysis of artery-waveform and gives nominal values. LiDCO is calibration with a small dose Lithium and gives absolute values. This study will examine relative changes, and calibration is not necessary.

The primary endpoints with respect to the hemodynamic effects of the interventions are group differences in systolic blood pressure and cardiac output the first 0-10 minutes after intervention. Secondary endpoints are other hemodynamic variables as stroke volume (SV), heart rate (HR), and systemic vascular resistance (SVR).

Demographic data and baseline measurements will be presented as mean (SD) if normally distributed or as median and range if not normally distributed, and group differences will be tested using the one-way ANOVA or Kruskal-Wallis tests, respectively. Baseline hemodynamic values represent measurements collected before administration of local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of cervical pre-cancer

Exclusion Criteria:

* Pregnancy
* Feeding mother
* Bad nutritional state
* Infection
* Treatment for hypertension
* Diabetes for many years or complications
* Cardiovascular disease
* Serious anemia
* Cardial arrythmia
* Serious liver-disease
* Hypersensitivity to local anesthesia of amide-type

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in Cardiac Output as measured by LiDCOplus monitor. | 0-10 minutes
  After paracervical Block.

SECONDARY OUTCOMES:
Changes in Stroke Volume as measured by LiDCOplus monitor. | 0-10 minutes
  After paracervical block.
Changes in Heart Rate as measured by LiDCOplus monitor. | 0-10 minutes
  After paracervical block.
Changes in Total Peripheral Resistance as measured by LiDCOplus monitor. | 0-10 minutes
  After paracervical Block.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Helge Sjøen, MD, Principal Investigator — Helse Fonna
Locations (1):
- Kirurgisk Klinikk-Anestesi, Haugesund, Rogaland, Norway

REFERENCES:
- [Background] Nesheim BI. Which local anesthetic is best suited for paracervical blocks? Acta Obstet Gynecol Scand. 1983;62(3):261-4. doi: 10.3109/00016348309155804. PMID 6353840
- [Background] Panda N, Verma RK, Panda NK. Efficacy and safety of high-concentration adrenaline wicks during functional endoscopic sinus surgery. J Otolaryngol Head Neck Surg. 2012 Apr;41(2):131-7. PMID 22569014
- [Background] Zhao F, Wang Z, Yang J, Sun J, Wang Q, Xu J. Low-dosage adrenaline induces transient marked decrease of blood pressure during functional endoscopic sinus surgery. Am J Rhinol. 2006 Mar-Apr;20(2):182-5. PMID 16686385 (Retraction: PMID 17181116 Am J Rhinol. 2006 Nov-Dec;20(6):673)
- [Background] Palomaki O, Huhtala H, Kirkinen P. A comparative study of the safety of 0.25% levobupivacaine and 0.25% racemic bupivacaine for paracervical block in the first stage of labor. Acta Obstet Gynecol Scand. 2005 Oct;84(10):956-61. doi: 10.1111/j.0001-6349.2005.00709.x. PMID 16167911
- [Background] Kerkkamp HE, Gielen MJ. Cardiovascular effects of epidural local anaesthetics. Comparison of 0.75% bupivacaine and 0.75% ropivacaine, both with adrenaline. Anaesthesia. 1991 May;46(5):361-5. doi: 10.1111/j.1365-2044.1991.tb09544.x. PMID 2035780
- [Background] de Leeuw MA, Slagt C, Hoeksema M, Zuurmond WW, Perez RS. Hemodynamic changes during a combined psoas compartment-sciatic nerve block for elective orthopedic surgery. Anesth Analg. 2011 Mar;112(3):719-24. doi: 10.1213/ANE.0b013e318206bc30. Epub 2010 Dec 14. PMID 21156977
- [Derived] Sjoeen GH, Falk RS, Hauge TH, Langesaeter E. Haemodynamic stability after paracervical block: A randomized, controlled, double-blind study comparing bupivacaine-adrenaline with bupivacaine. Acta Anaesthesiol Scand. 2019 Mar;63(3):373-380. doi: 10.1111/aas.13259. Epub 2018 Sep 10. PMID 30203440